CLINICAL TRIAL: NCT00486421
Title: A Pilot Study of Rituximab in Combination With Corticosteroids for the Initial Treatment of Immune Thrombocytopenic Purpura
Brief Title: Rituximab and Prednisone as First-Line Therapy in Treating Patients With Immune Thrombocytopenic Purpura
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000529883; P30CA015083 (NIH); MC0481 (Other: Mayo Clinic Cancer Center); 2071-04 (Other: Mayo Clinic IRB); U2985s (Other: Genentech protocol)
Record Dates: First submitted 2007-06-13; First posted 2007-06-14 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2014-10

CONDITIONS: Nonneoplastic Condition
Keywords: idiopathic thrombocytopenic purpura
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Rituximab; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PRED & RITUX (Experimental)
  Interventions: Biological: Rituximab; Drug: Prednisone

INTERVENTIONS:
Biological: Rituximab — 375mg/m2 IV weekly times 4 (days 1, 8, 15, 22)
  Other Names: Rituxan
Drug: Prednisone — 1mg/kg/d PO, taper to off by 8 weeks

SUMMARY:
RATIONALE: Rituximab and prednisone may increase the number of platelets in patients with immune thrombocytopenic purpura.

PURPOSE: This phase II trial is studying the side effects and how well giving rituximab together with prednisone works as first-line therapy in treating patients with immune thrombocytopenic purpura.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of rituximab, when administered with standard prednisone treatment, in maintaining a platelet count ≥ 50,000/mm³ at 6 months without further therapies (e.g., splenectomy or other salvage therapies) in patients with immune thrombocytopenic purpura.
* Determine the safety of this regimen in these patients.

Secondary

* Determine the time to platelet recovery in patients treated with this regimen.
* Determine the duration of platelet recovery in patients treated with this regimen.
* Assess efficacy of this regimen in preventing spontaneous bleeding events in these patients.
* Determine the response in patients treated with this regimen.

OUTLINE: This is a pilot study.

Patients receive rituximab IV on days 1, 8, 15, and 22 and oral prednisone once daily on days 1-14 followed by a taper to day 56. Treatment is administered in the absence of disease relapse or unacceptable toxicity.

After completion of study therapy, patients are followed periodically for up to 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of immune thrombocytopenic purpura (ITP)

  * Diagnosis must be made according to American Society of Hematology diagnostic guidelines by a member of Mayo Rochester's Division of Hematology/Oncology within the past year
  * ITP must be confirmed by bone marrow aspiration and biopsy in all patients ≥ 60 years of age*

    * Bone marrow studies performed outside Mayo must be reviewed by a Mayo hematopathologist to confirm diagnosis and exclude evidence of other hematologic disorders NOTE: *Bone marrow evaluation is discretionary for all other patients
* Requires treatment, as defined by 1 of the following parameters:

  * Platelet count ≤ 30,000/mm³
  * Platelet count ≤ 50,000/mm³ with episodic bleeding (i.e., spontaneous or with minimal trauma) requiring treatment
* No concurrent diagnosis of a condition known to cause secondary immune (or nonimmune) thrombocytopenia, including, but not limited to, any of the following:

  * Rheumatological conditions, such as lupus, rheumatoid arthritis, scleroderma, or mixed connective tissue disorder

    * Patients with positive serologies and no concurrent, clinically evident condition are eligible
  * HIV positive or AIDS
  * Non-Hodgkin's lymphoma, Hodgkin's lymphoma, chronic lymphocytic lymphoma, multiple myeloma, or other malignant hematological conditions
  * Clinically evident antiphospholipid antibody syndrome* or heparin-induced thrombocytopenia
  * Clinically overt liver disease, hepatitis B surface antigen positive, hepatitis C serology positive, or evidence of a microangiopathic hemolytic anemia, such as disseminated intravascular coagulation, hemolytic-uremic syndrome, thrombotic thrombocytopenic purpura, or preeclampsia NOTE: *Positive laboratory tests without the defined clinical criteria for a diagnosis of antiphospholipid antibody syndrome is allowed

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Creatinine ≤ 2 times upper limit of normal (ULN)
* Direct bilirubin ≤ 1.5 times ULN
* Total bilirubin ≤ 1.5 times ULN
* AST ≤ 2.5 times ULN
* Hemoglobin ≥ 10 g/dL
* WBC ≥ 3,000/mm³
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No hypersensitivity to murine or chimeric proteins
* No other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk for treatment complications
* Able to take a proton-pump inhibitor while on corticosteroids
* No unresolved or incompletely treated infection within the past 14 days

PRIOR CONCURRENT THERAPY:

* No prior corticosteroid therapy since the diagnosis of ITP

  * Corticosteroid therapy is allowed for up to 14 days prior to study entry, once the baseline CBC has been established
* No prior rituximab
* No other concurrent therapy for ITP, including androgens, IV immunoglobulins, RH_o (D) immune globulin, cyclosporine, or azathioprine sodium

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2007-01; Primary Completion 2008-05 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Failure-free survival at 6 months | 6 months

SECONDARY OUTCOMES:
Time to platelet recovery | 1 year
Duration of platelet recovery | 1 year
Effect of treatment on prevention of spontaneous bleeding events | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ruben A. Mesa, M.D., Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States